CLINICAL TRIAL: NCT05479643
Title: A Pilot Study for a Novel and Personalized Voice Restoration Device for Patients With Laryngectomy
Brief Title: A Personalized Voice Restoration Device for Patients With Laryngectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-03024627
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Dysphonia; Aphonia
MeSH Terms: conditions — Dysphonia; Aphonia | interventions — Electromyography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Patients with Aphonia or Dysphonia (Experimental): Participants with Aphonia or Dysphonia will be asked to recite phrases with sEMG attached to articulatory muscles.
  Interventions: Device: Surface Electromyography
- Healthy Volunteers (Placebo Comparator): Healthy Volunteer will be asked to recite phrases with sEMG attached to articulatory muscles.
  Interventions: Device: Surface Electromyography

INTERVENTIONS:
Device: Surface Electromyography — Surface ElectroMyoGraphy (SEMG) is a non-invasive technique for measuring muscle electrical activity that occurs during muscle contraction and relaxation cycles. Electrodes will be attached with a AgCl gel to muscles used for articulation.

SUMMARY:
The investigators will conduct a pilot experiment for a novel and personalized method for voice restoration using machine learning applied to surface EMG (sEMG) signal from articulatory muscles of the face and the neck allowing recognition of silent speech. The investigators predict that the use novel personalized method for voice restoration will be feasible and successful for patients.

DETAILED DESCRIPTION:
This is a prospective pilot study evaluating the feasibility of a personalized voice restoration device and patients' experience with it. Study participation will include a one-time visit where subjects will read passages and phrases. Acoustic and signal data will be captured. Machine learning will be applied to the data to classify words. Subjects will also participate in a qualitative interview about their experience with voice restoration devices.

ELIGIBILITY:
Inclusion Criteria:

Group A: Healthy Volunteers

1. Adult subjects, 18 or older
2. Without any voice impairments

Group B: Subjects with Aphonia or Dysphonia

1. Adult subjects, 18 or older
2. Documentation of severe dysphonia and/or aphonia, or a GRBAS score > 0 (GRBAS is a scale that can be used to assess voice quality of subjects who do not have a recorded history of dysphonia or aphonia. The GRBAS scale evaluates for grade, roughness, breathiness, asthenia, and strain).

Exclusion Criteria:

- Group A: Healthy Volunteers

1. Voice impairment

Group B: Subjects with Aphonia or Dysphonia

1. Subjects whose face muscles are entirely paralyzed

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2027-12-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Words and Numbers Correctly Identified | "During Procedure/use of Surface ElectroMyoGraphy"
  Accuracy of sEMG signal will be determined by subjects reciting common phrases. Subjects will recite the "Rainbow Passage" 10 times. Subjects will be asked to count from 1-10 once. Subjects will recite the alphabet once.
Subject experience with voice restoration devices: Qualitative | 10 minutes after the time of intervention
  Subject will be asked to complete a semi-structured interview about their experience with voice restoration devices. Categories of response include voice/communication history, experience with previous voice restoration devices, experience with our device, and suggestions for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs Rameau, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No